CLINICAL TRIAL: NCT02729805
Title: Effects of Intraoperative Intravenous Ketamine on Chronic Pain After Mastectomy
Brief Title: Intraoperative Ketamine on Chronic Pain After Mastectomy
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW15-079
Record Dates: First submitted 2015-06-28; First posted 2016-04-06 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: ketamine; chronic pain; mastectomy; acute pain
MeSH Terms: conditions — Chronic Pain; Acute Pain | interventions — Sodium Chloride; Control Groups; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (Placebo Comparator): A syringe of 50 ml 0.9% normal saline will be prepared as placebo for infusion and a syringe of 10ml 0.9% normal saline for bolus injection.
  Interventions: Drug: Saline
- Ketamine 0.5mg/kg (Active Comparator): A bolus injection of intravenous ketamine at a dose of 0.5mg/kg during anaesthetic induction before skin incision followed by 0.25mg/kg/hr intravenous ketamine infusion during the operation.
  Interventions: Drug: Ketamine 0.5mg/kg
- Ketamine 0.75mg/kg (Experimental): A bolus injection of intravenous ketamine at a dose of 0.75mg/kg during anaesthetic induction before skin incision followed by 0.5mg/kg/hr intravenous ketamine infusion during the operation.
  Interventions: Drug: Ketamine 0.75mg/kg

INTERVENTIONS:
Drug: Saline — 10ml bolus injection of saline followed by intravenous infusion of saline during the operation
  Other Names: Control group
  Arms: Saline
Drug: Ketamine 0.5mg/kg — 0.5mg/kg intravenous ketamine injection followed by 0.25mg/kg/hr intravenous ketamine infusion during the operation
  Other Names: Group K1
  Arms: Ketamine 0.5mg/kg
Drug: Ketamine 0.75mg/kg — 0.75mg/kg intravenous ketamine injection followed by 0.5mg/kg/hr intravenous ketamine infusion during the operation
  Other Names: Group K2
  Arms: Ketamine 0.75mg/kg

SUMMARY:
Preventive analgesia is when an administered analgesic drug provides reduction in pain beyond its duration of action. This can be used to reduce acute postoperative pain and prevent occurrence of chronic post-surgical pain.

According to the International Association for the Study of Pain (IASP), chronic pain can be defined as pain that persisted beyond the time of normal tissue healing (usually 3 months) and that was not related to other causes. Mastectomy is associated with a high incidence of chronic post-surgical pain. Breast cancer is the most common malignancy affecting females around the world. Many undergo mastectomy as part of curative treatment. However, a significant proportion of patients experience chronic post-surgical pain. This results in significant negative impact on physical, psychological and social wellbeing.

Ketamine is an intravenous anaesthetic drug with analgesic effects. It can be used to treat both acute and chronic pain. A recent meta-analysis of different surgeries showed that patients receiving ketamine had a modest but statistically significant reduction in incidence of chronic post-surgical pain. In a small sample single dose pilot study, patients given low dose intravenous ketamine intraoperatively had a statistically non-significant reduction in incidence of pain around the surgical scar at three months after radical mastectomy. Randomized control trials with larger sample sizes are needed to determine the effectiveness and optimal dosing regime of ketamine for reduction of chronic post-mastectomy pain. It is therefore hypothesized that intravenous ketamine given intraoperatively will reduce the incidence and severity of chronic pain after modified radical mastectomy. A double blind randomized controlled trial comparing placebo group with two different doses of ketamine is proposed.

The mechanism of action of ketamine in reducing pain is complex and multiple. How ketamine can prevent and reduce chronic pain is unknown. Ketamine has been shown to reduce immediate gene expression at site of mechanical injury. Transient Receptor Potential Vanilloid 1 (TRPV1) and Transient Receptor Ankyrin 1 (TRPA1) are receptors shown to mediate acute and chronic pain. Ketamine, shown to affect gene expression, may alter the expression of TRPV1 and TRPA1 via epigenetic mechanisms.

DETAILED DESCRIPTION:
Procedures Patients will be approached at the preadmission clinic or in the general ward before operation. The analgesic methods will be explained and s/he will be recruited into the study if s/he agrees. The patient will be randomized into one of three groups. The patients in the first group (C) will receive intraoperative morphine, local wound infiltration with local anaesthetic, cyclooxygenase-2 (COX-2) inhibitor post-operatively, and post operative Patient Controlled Analgesia (PCA) morphine. Patients in the second (K1) and third groups (K2) will receive different doses of intraoperative intravenous ketamine in addition to intraoperative morphine, local wound infiltration with local anaesthetic, COX-2 inhibitor, and PCA morphine.

Randomization and blinding Patients recruited for mastectomy will be stratified in randomization. To ensure equal distribution of patients between each type of operation (modified radical mastectomy with axillary dissection and mastectomy with sentinel lymph node without axillary dissection) block randomization will be used. There will be 9 blocks of 15 patients for each type of operation. The allocation order will be selected by a computer generated random sequence.

This is a double blind randomized control trial. Both the patients and the investigators will be blinded to the allocated analgesic modalities: ie the administration of ketamine. Ketamine or normal saline (placebo) will be prepared by clinical staff who will not participate in observation and data analysis.

Data collection

The following data will be collected during the perioperative period:

* Demographics
* Time of admission
* Intraoperative vital signs (blood pressure, heart rate, oxygen saturation)
* Estimated intraoperative blood loss
* Volume of intraoperative fluid/blood infusion
* Duration of anaesthetic or analgesic procedures before surgical procedure
* Duration of surgical procedures
* Time from end of surgical procedure to extubation
* Demands and goods of PCA morphine use
* Cumulative morphine consumption
* Vital signs and NRS pain scores at rest and during cough/ipsilateral arm movement upon recovery every hour for 4 hours, and then once every 4 hours for up to 5 days during the time that PCA morphine is used. Afterwards, these data will be collected daily until discharge
* Dose and frequency of rescues analgesics (Intra muscular injection of morphine) used
* Side effects of analgesics (pruritus, dizziness, nausea, vomiting, psychomimetic effects etc.)
* Time to recovery of food intake (fluid, semisolid and solid diet)
* Time to ambulation (bed rest, sit up, sit out of bed, walk with aid, walk without aid)
* Surgical and anaesthetic complications, if any (wound infection, urinary retention, etc.)
* Time to discharge
* Patient satisfaction upon discharge

The following data would be obtained at 3 and 6 months after surgery:

* The presence of chronic pain
* The location of pain
* Pain severity (Numerical Rating scale (NRS) score): at rest, during cough/movement of the ipsilateral arm
* Any analgesic consumption
* Nature of pain: nociceptive, neuropathic
* Timing of pain occurrence: continuous, related to movement, intermittent.
* Any abnormal sensation or loss of sensation over operated side.
* Health related quality of life (HRQOL) data obtained with the Chinese (Hong Kong) version of Short Form-12 version 2 (SF12v2) Health Survey.
* Patient's psychological condition will be assessed with the Hospital Anxiety and Depression Scale (HADS) questionnaire.
* Physical examination to check for any brush allodynia and pinprick hyperalgesia

Other data:

* Survival status at 6 and 12 months after operation
* Any recurrence of disease
* Treatment with radiotherapy or chemotherapy
* If, at certain time point after operation, patient cannot be managed according to the protocol due to any reason such as development of complication, no further data will be collected.

Blood taking for assessment of genetic, epigenetic factors and biomarkers Blood (10mls in tubes with Ethylenediaminetetraacetic acid (EDTA) as preservative) will be taken immediately pre-surgery, immediately post-surgery, one day post-surgery, three days post-surgery, and at 3 and 6-months after surgery.

Data analysis Intention-to-treat will be used. Patients will remain in their initial designated groups for data analysis even if there is a change in surgical or anaesthetic/analgesic management, as long as they have had a laparoscopic incision during the operation.

Statistical methods used:

* Incidence of chronic post mastectomy pain: Chi-Square test
* NRS pain scores at 3 and 6 months after surgery, estimated blood loss, duration of anaesthetic, analgesic and surgical procedures, time to extubation, tries and goods of PCA morphine used, cumulative morphine consumption, dose and frequency of rescue analgesic used, time to food intake and ambulation, time to discharge, patient satisfaction: Kruskal-Wallis test
* Acute NRS pain scores over 48 hours: Expressed as area under the curve (AUC) using the trapezoid rule and compared using Kruskal-Wallis test.
* Patient demographic data: One way Analysis of Variance (ANOVA) and chi-square test.
* Intraoperative vital signs, HRQOL, HADS: Repeated measures ANOVA (with Bonferroni correction when appropriate)
* Side effects and postoperative complications: Chi Square test
* Binary logistic regression will be used to assess the relationship between development (or non-development) of chronic pain and DNA methylation status of TRPV1 and TRPA1.
* When a significant result was obtained, t-test or Mann-Whitney test for numerical values and Chi-square test for categorical data will be applied for post hoc pairwise comparisons.

ELIGIBILITY:
Inclusion Criteria:

* the American Society of Anesthesiologists adopted physical status classification system (ASA) I-III
* Age 18-80 years old
* Scheduled for 1) modified radical mastectomy (including axillary lymph node dissection) and 2) mastectomy with sentinel lymph node (without axillary dissection). These are the common surgical treatments for breast cancer.

Exclusion Criteria:

* Radical mastectomy, wide local excision or lumpectomy
* Known allergy to opioids, local anaesthetic drugs, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors
* History of chronic pain
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120 micromol/L
* Pre-existing neurological or muscular disorders
* Psychiatric illness
* Impaired or retarded mental state
* Not self ambulatory before operation
* Difficulties in using patient controlled analgesia (PCA)
* Pregnancy
* Local infection
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2015-08-18 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Severity of chronic pain | At postoperative 3 months
  Determine the severity using numerical rating scale

SECONDARY OUTCOMES:
Incidence of neuropathic pain | At postoperative 3 months
  Determine the incidence of neuropathic pain using Identification Pain Questionnaire for Neuropathic Pain (ID-NeP)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided